CLINICAL TRIAL: NCT05509127
Title: Evaluation of Cervical Restorations Performance Using Modified Universal Adhesive Compared to Conventional Universal Adhesive: A Randomized Clinical Trial
Brief Title: Evaluation of Cervical Restorations Performance Using Modified Universal Adhesive
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Gamal Dawoud, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Modified Universal Adhesive
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Clinical Performance
Keywords: Performance; Carious; Cervical; Universal adhesive; USPHS criteria
MeSH Terms: interventions — Adhesives

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carious cervical lesions treated with modified universal adhesive (Experimental): Preparation of class V cavity with removal of caries and beveling of margins is done followed by total etching prior to application of modified universal adhesive. The cavity is then restored with nano-filled resin composite.
  Interventions: Drug: Modified universal adhesive
- Carious cervical lesions treated with conventional universal adhesive (Active Comparator): Preparation of class V cavity with removal of caries and beveling of margins is done followed by total etching prior to application of conventional universal adhesive. The cavity is then restored with nano-filled resin composite.
  Interventions: Drug: Conventional universal adhesive

INTERVENTIONS:
Drug: Modified universal adhesive — Application of the modified universal adhesive is done according to manufacturer's instructions using a micro-brush. It is actively rubbed for 20 seconds, gently air-dried for 5 seconds then light cured for 20 seconds.
  Other Names: 3M ESPE™ Scotchbond Universal Plus Adhesive
  Arms: Carious cervical lesions treated with modified universal adhesive
Drug: Conventional universal adhesive — Application of the conventional Single Bond Universal adhesive is done using a micro-brush followed by rubbing for 20 seconds, gentle air drying for 5 seconds then light curing for 20 seconds.
  Other Names: 3M ESPE™ Single Bond Universal Adhesive
  Arms: Carious cervical lesions treated with conventional universal adhesive

SUMMARY:
Class V restorations are evaluated to reveal whether the use of modified universal adhesive will have a similar performance compared to conventional universal adhesive or not.

DETAILED DESCRIPTION:
The innovative Scotchbond Universal Plus Adhesive offers all the benefits of its predecessor, Single Bond Universal Adhesive as demonstrated by a 3M field evaluation comparing the performance of the two products. These benefits include:

* Compatibility with all etching techniques - total-etch, self-etch, and selective enamel etch.
* Usage with direct and indirect indications.
* Bonding to all dental surfaces without the need for separate primers or silanes
* Virtually no post-operative sensitivity.

The newly modified adhesive with its careful formulation offers:

* Radiopacity like dentin to reduce the risk of X-ray misdiagnosis and overtreatment.
* Ability to bond and seal caries-affected dentin to support minimally invasive preparation guidelines and maximize preservation of natural tooth structure.
* Adhesion to all dental substrates and all direct and indirect materials, including glass ceramics.
* Full dual- and self-cure compatibility without the need for an additional dual-cure activator bottle.
* A BPA derivative-free formulation to alleviate concerns about BPA in dental materials
* A fully aligned system with RelyX™ Universal Resin Cement, offering excellent bond strength for virtually all dual-cure resin cement indications.

As with any new material or technique, long-term clinical evaluations are needed to demonstrate the value of universal bonding agents adequately. So, the aim of this study is to evaluate the clinical performance of the modified universal adhesive, versus the conventional universal adhesive, for restoring carious class V cavities over one year and a half.

ELIGIBILITY:
Inclusion Criteria:

* Small to moderate carious cervical lesions. (ICDAS scores 3,4)
* Upper premolar teeth.
* Good oral hygiene (mild to moderate plaque accumulation)
* Vital teeth with no signs of irreversible pulpitis.
* Presence of favorable occlusion and normal contact with adjacent teeth.

Exclusion Criteria:

* Patients with systemic diseases, severe medical complications or allergic history concerning methacrylates.
* Lack of patient compliance, pregnancy, rampant caries, heavy smoking or xerostomia.
* Evidence of parafunctional habits and TMJ disorders.
* Class V lesions in molars.
* Non-carious cervical lesions.
* Deep carious defects (close to pulp, less than 1 mm distance).
* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Endodontically treated teeth.
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism.
* Severe periodontal affection.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Marginal adaptation | Baseline, 6 months, 12 months, 18 months and 24 months.
  using Modified USPHS criteria

SECONDARY OUTCOMES:
Marginal discoloration | Baseline, 6 months, 12 months, 18 months and 24 months.
  using Modified USPHS criteria
Post-operative sensitivity | Baseline, 6 months, 12 months, 18 months and 24 months.
  using Modified USPHS criteria
Retention | Baseline, 6 months, 12 months, 18 months and 24 months.
  using Modified USPHS criteria
Secondary caries | Baseline, 6 months, 12 months, 18 months and 24 months.
  using Modified USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt